CLINICAL TRIAL: NCT04029311
Title: Comparison of Two Techniques of Combination Therapy for Treatment of Obstructive Sleep Apnea (OSA)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Joseph Adame (Individual)
Responsible Party: Sponsor-Investigator, Joseph Adame, J. Michael Adame, DDS, Principal Investigator, Adame, J. Michael, D.D.S.
Organization: Adame, J. Michael, D.D.S. (Individual)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20170991
Record Dates: First submitted 2019-07-19; First posted 2019-07-23 (Actual); Results first posted 2021-04-02 (Actual); Last update posted 2021-04-02 (Actual); Status verified 2021-03

CONDITIONS: Treatment for Obstructive Sleep Apnea

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Combination Therapy with Preferred Mask (Experimental): Preferred Mask refers to a type of existing medical mask used for PAP therapy.
  Interventions: Device: Nuance Pro; Device: autoPAP
- Combination Therapy with Custom Mask (Experimental): Custom Mask refers to a mask which is supported by an interface which attaches directly to the patient's oral appliance.
  Interventions: Device: autoPAP; Device: TAP PAP

INTERVENTIONS:
Device: Nuance Pro — Study compares Nuance Pro plus Automatic Positive Airway Pressure (autoPAP) vs TAP PAP plus autoPAP
  Other Names: TAP PAP
  Arms: Combination Therapy with Preferred Mask
Device: autoPAP — autoPAP
Device: TAP PAP — TAP PAP
  Arms: Combination Therapy with Custom Mask

SUMMARY:
To study the effects of two combination therapies for patients with obstructive sleep apnea (OSA) who have been both intolerant to Positive Airway Pressure (PAP) therapy and sub-therapeutic to oral appliance therapy.

Hypothesis

1. There is a difference between Continuous Positive Airway Pressure (CPAP) vs CPAP/Oral Appliance (OA) connect vs CPAP/OA disconnected in terms of:

1. Apnea Hypopnea Index (AHI) reduction
2. Amount of side effects
3. Amount of Leaks
4. Hours of use (compliance)
5. CPAP pressure

2. There is a difference between connected and disconnected for the following symptoms:

1. Epworth sleepiness Scale (ESS)
2. Functional Outcomes of Sleep Questionnaire (FOSQ)
3. Side effects Study Design - randomized prospective parallel

ELIGIBILITY:
Inclusion Criteria: Baseline diagnosis AHI > or = 5 plus ESS . or = 10.

* PAP Intolerance
* Partial Response to oral appliance therapy: AHI > 5
* Age: > 18 Exclusion Criteria: History of daily use of alcohol, narcotics or Central Nervous System (CNS) depressants.
* Diagnosis of Central Sleep Apnea
* Pregnancy
* Edentulous
* Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2017-06-08 (Actual); Primary Completion 2019-02-06 (Actual); Study Completion 2019-05-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- J. Michael Adame, DDS, PA, Edinburg, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Combination Therapy With Preferred Mask: Preferred Mask refers to a type of existing medical mask used for Positive Airway Pressure (PAP) therapy.
  Nuance Pro: Study compares Nuance Pro plus Automatic Positive Airway (autoPAP ) vs TAP PAP plus autoPAP
  autoPAP: autoPAP
Period: Overall Study
Arm/Group | Combination Therapy With Preferred Mask | Combination Therapy With Custom Mask
Started | 15 | 13
Completed | 12 | 13
Not Completed | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Combination Therapy With Preferred Mask: Preferred Mask refers to a type of existing medical mask used for PAP therapy.
  Nuance Pro: Study compares Nuance Pro plus autoPAP vs TAP PAP plus autoPAP
  autoPAP: autoPAP
- Total: Total of all reporting groups
Arm/Group | Combination Therapy With Preferred Mask | Combination Therapy With Custom Mask | Total
Number analyzed (Participants) | 15 | 13 | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 11 | 20
  >=65 years | 6 | 2 | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.9 (12.7) | 54.5 (8.6) | 56.3 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 6 | 15
  Male | 6 | 7 | 13
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 15 | 13 | 28
BMI [Mean (Standard Deviation); unit: kg/m^2] | 34.4 (8.4) | 32.9 (7.5) | 33.8 (7.9)

OUTCOME MEASURES:

1. Primary Outcome: Apnea-Hypopnea Index
Description: Episodes per hour that the patient experiences apneas and/or hypopneas
Time Frame: 2 months
Population: Missing data from 1 participant in Combination Therapy with Preferred Mask group
Measure: Mean (Standard Deviation); unit: episodes/hour
Arm/Group | Combination Therapy With Preferred Mask | Combination Therapy With Custom Mask
Number analyzed (Participants) | 11 | 13
episodes/hour | 4.1 (3.6) | 3.6 (2.7)

2. Primary Outcome: PAP Pressure
Description: The pressure required to treat the patient successfully
Time Frame: 2 months
Population: Missing data from 1 participant in Combination Therapy with Preferred Mask group.
Measure: Mean (Standard Deviation); unit: cmH2O
Arm/Group | Combination Therapy With Preferred Mask | Combination Therapy With Custom Mask
Number analyzed (Participants) | 11 | 13
cmH2O | 9.6 (1.8) | 8.6 (1.9)

3. Primary Outcome: Leaks
Description: The Liters/Minute of leaking of the PAP machine
Time Frame: 2 months
Population: Missing data from 1 participant in Combination Therapy with Preferred Mask group.
Measure: Mean (Standard Deviation); unit: L/min
Arm/Group | Combination Therapy With Preferred Mask | Combination Therapy With Custom Mask
Number analyzed (Participants) | 11 | 13
L/min | 15.1 (8.0) | 16.7 (14.1)

4. Primary Outcome: Hours of Use
Description: The average hours of use per night of each of the combination therapies
Time Frame: 2 months
Population: Missing data from 1 participant in Combination Therapy with Preferred Mask group.
Measure: Mean (Standard Deviation); unit: hours per night
Arm/Group | Combination Therapy With Preferred Mask | Combination Therapy With Custom Mask
Number analyzed (Participants) | 11 | 13
hours per night | 6.0 (1.9) | 5.9 (2.4)

5. Primary Outcome: Epworth Sleepiness Scale (ESS)
Description: The ESS is a self-administered questionnaire with 8 questions. The score can range from 0 to 24. The higher the ESS score, the higher that person's average sleep propensity in daily life.
Time Frame: 2 months
Population: Missing data from 1 participant in Combination Therapy with Preferred Mask group.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Combination Therapy With Preferred Mask | Combination Therapy With Custom Mask
Number analyzed (Participants) | 11 | 13
score on a scale | 5.5 (4.0) | 5.8 (2.7)

6. Primary Outcome: Functional Outcomes Sleep Questionnaire (FOSQ)
Description: FOSQ is a disease specific quality of life questionnaire to determine how sleepiness interferes one's quality of life. The total score range from 5 to 20 (10 questions, 1-4 points per each). The lower values represent a worse quality of life.
Time Frame: 2 months
Population: Missing data from 1 participant in Combination Therapy with Preferred Mask group.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Combination Therapy With Preferred Mask | Combination Therapy With Custom Mask
Number analyzed (Participants) | 11 | 13
score on a scale | 36.3 (3.8) | 36.2 (2.8)

7. Primary Outcome: Intolerance Questionnaire
Description: This questionnaire consists of 4 questions to determine the frequency of 4 typical side-effects from positive airway pressure therapy. The score ranges from 0 to 16 (4 questions, 0-4 points per each). The higher value represent worse side effects.
Time Frame: 2 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Combination Therapy With Preferred Mask | Combination Therapy With Custom Mask
Number analyzed (Participants) | 11 | 13
score on a scale | 2.7 (2.4) | 3.4 (2.7)

ADVERSE EVENTS:
Time Frame: 2 months
Arm/Group | Combination Therapy With Preferred Mask | Combination Therapy With Custom Mask
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/13
Other Adverse Events (participants affected / at risk) | 0/15 | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2015-06-16): https://cdn.clinicaltrials.gov/large-docs/11/NCT04029311/Prot_SAP_ICF_001.pdf